CLINICAL TRIAL: NCT01546506
Title: Confirmation of the Antiviral Effects of Midodrine Identified With a Gene Expression Signature-based Screening of Inluenza A Virus Infected Cells
Acronym: FLUMED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010.654/58
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Influenza A Virus Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midodrine (Experimental): Midodrine 2.5 mg orally 3 times daily, 5 day-treatment.
  Interventions: Drug: Gutron® treatment
- No treatment (No Intervention)

INTERVENTIONS:
Drug: Gutron® treatment — Midodrine 2.5 mg orally 3 times daily, 5 day-treatment.
  Arms: Midodrine

SUMMARY:
Rationale:

Classical antiviral therapies target viral proteins and are consequently subject to resistance. To counteract this limitation, alternative strategies have been developed that target cellular factors. We hypothesized that such an approach could also be useful to identify broad-spectrum antivirals. The influenza A virus was used as a model for its viral diversity and because of the need to develop therapies against unpredictable viruses as recently underlined by the H1N1 pandemic. Gene-expression signature-based screening identified broadly effective influenza A antivirals. Midodrine showed great results in inhibiting viral growth and was the most suited to confirm its efficacy in vivo.

The main objective of the study is to assess the efficacy of midodrine taken at usual recommended dose (7.5mg/day) versus no treatment on viral replication kinetics of virus Influenza A.

Secondary objectives: evaluation of the number of patients with a normalized viral load 2, 3 5 and 7 days post-treatment; description of the anti-viral efficacy of midodrine defined as the delay to obtain a prolonged negativity of viral RNA; description of the tolerance of midodrine, evaluation of the clinical response to study treatment; evaluation of the dynamic of viral replication; analysis of the frequency of emergence of mutants and associated resistance.

Methods:

This is a multicenter, randomized, open-label study comparing patients aged 18 to 65 years infected by influenza A virus. Nasopharyngeal washing will be performed at day 0 (randomization), 2, 3, 5 to show the viral replication evolution.

161 patients will be randomized as follows :

* Arm 1 : Midodrine, 2.5 mg, 3 times a day
* Arm 2 : No treatment The recruitment is performed by general practitioners in the Lyon area.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18 to 65 years,
* with no long-term illness,
* presenting flu-like symptoms for less than 42 hours (nasal congestion, sore throat, muscle soreness, asthenia, headache, chills/sweating, fever…),
* infection with influenza A virus confirmed with a quick diagnostic test,
* outpatient care,
* must provide signed and informed consent,
* beneficiary of a health insurance.

Exclusion Criteria:

* severe form of flu,
* pregnant women or positive pregnancy test,
* breastfeeding women,
* women of childbearing-potential with no efficient contraceptive,
* history of chronic respiratory disease : asthma or chronic obstructive pulmonary disease,
* renal failure,
* Raynaud's disease,
* history of epilepsy, confusion, hallucinations or of psychoneurotic state,
* patients with an increased cardiovascular risk (> 20% according to the Framingham scale) or with a cardiovascular history,
* patients having a congestive heart failure, swollen legs or a posture hypotension,
* patients who received a influenza vaccine for seasons 2011-2012 or 2012-2013,
* known hypersensitivity to any component of the treatment,
* topical use of nasal decongestant (except physiological serum),
* use of steroids, immunosuppressive or antipsychotics drugs (including treatments for nausea),
* use of indirect sympathomimetics drugs (ephedrine, methylphenidate, phenylephrine, pseudoephedrine),
* use of dopaminergic ergot alkaloids (bromocriptine, cabergoline, lisuride, pergolide) or vasoconstrictor ergot alkaloids (dihydroergotamine, ergotamine, methylergométrine, methylsergide),
* known hypertension treated or not,
* history of bradycardia,
* history of urinary retention,
* severe cardiopathy,
* acute angle-closure glaucoma,
* severe obliterative vasculopathy,
* vasospasm,
* thyrotoxicosis,
* pheochromocytoma,
* history of angina pectoris,
* use of guanethidine and related, iproniazide (non selective MAOIs), alpha-blockers and digitalis drugs
* use of neuraminidase inhibitors: oseltamivir, zanamivir; and M2 proton-selective ion channel inhibitors: amantadine and rimantadine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Comparison of viral replication kinetics between the 2 arms | 7 days
  Comparison of the viral load slopes for 7 days post-study treatment start. Viral load will be measured at day 0, 2, 3, 5, and 7

SECONDARY OUTCOMES:
Percentage of patients with a normalized viral load | 7 days
  A normal viral load is defined as a value below the positive threshold of 3 in RT-qPCR at day 2, 3, 5 and 7
Duration and severity of flu symptoms | 7 days
Frequency, duration and level of replication of the virus in nose samples | 7 days
Viral resistance and decrease of sensitivity of collected strains | 7 days
Tolerance of midodrine : incidence of adverse effects | 7 days
  Side effects will be checked at each visit and reported for the entire study timeframe.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno LINA, MD, PhD, Principal Investigator — Laboratoire de virologie, Institut de microbiologie, Centre de Biologie et de Pathologie EST, Groupement Hospitalier Est, Hospices Civils de Lyon
Locations (39):
- France (39):
  - Cabinet Médical du Dr ALIBERT, Bron
  - Cabinet Médical du Dr CURE, Bron
  - Centre d'Investigation Clinique de Lyon, Bron
  - Cabinet du Dr DAHAN, Decine Charpieu
  - Cabinet du Dr MADELON, Décine Charpieu
  - Cabinet Médical du Dr HILLION, Lyon
  - Cabient Médical du Dr PIOS, Lyon
  - Cabinet du Dr ATTALI, Lyon
  - Cabinet du Dr COUTY, Lyon
  - Hôpital D'Instruction des Armées Desgenettes, Lyon
  - Cabinet Médical du Dr FORGEOIS, Lyon
  - Cabinet Médical du Dr TERRASSE, Lyon
  - Cabinet du Dr THIBAUT, Lyon
  - Cabinet Médical du Dr BUGEL, Lyon
  - Cabinet Médical du Dr CHAPDANIEL, Lyon
  - Cabinet du Dr AKIKI, Lyon
  - Cabinet du Dr BOURAS, Lyon
  - Cabinet du Dr GREVE, Lyon
  - Cabinet du Dr MANOELIAN, Lyon
  - Cabinet du Dr ROCHE, Lyon
  - Cabinet du Dr AZULAY TEBOUL, Lyon
  - Cabinet du Dr DRUT, Lyon
  - Cabinet Médical du Dr SAINT-OLIVE, Lyon
  - Cabinet du Dr JACQUET, Meyzieu
  - Cabinet du Dr FARHAT, Saint-Pierre-de-Chandieu
  - Cabinet du Dr CHAMPETIER, Saint-Priest
  - Cabinet Médical du Dr SMIT, Saint-Priest
  - Cbinet Médical du Dr CEZANNE-BERT, Saint-Priest
  - Cabinet Médical du Dr DUBOIS, Saint-Symphorien-dOzon
  - Cabinet du Dr CHAIZE, Vénissieux
  - Cabinet Médical du Dr MARTIN, Vénissieux
  - Cabinet Médical du Dr THEOULE, Vénissieux
  - Cabinet Médical du Dr MOREAU, Villefontaine
  - Cabinet Médical du Dr BUFFLER, Villeurbanne
  - Cabinet Médical du Dr KESSOUS, Villeurbanne
  - Cabinet Médical du Dr MONLOUBOU, Villeurbanne
  - Cabinet Médical du Dr PERDRIX, Villeurbanne
  - Cabinet Médical du Dr PILLARS, Villeurbanne
  - Cabinet Médical du Dr WEBER, Villeurbanne